CLINICAL TRIAL: NCT06067269
Title: High Precision Stereotactic Radiotherapy to the Whole Prostate With Focal Boost and Varying Hormonal Therapy (HEATWAVE)
Brief Title: Hormone Therapy (Apalutamide) and Image-guided Stereotactic Body Radiation Therapy for the Treatment of Patients With Prostate Cancer, HEATWAVE Trial
Acronym: HEATWAVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-000429; NCI-2023-06647 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-09-21; First posted 2023-10-04 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Prostate Adenocarcinoma; Stage II Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Specimen Handling; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (apalutamide, SBRT) (Experimental): Patients receive apalutamide PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 or 12 months in the absence of disease progression or unacceptable toxicity. Patients undergo SBRT for 5 fractions over 1-2 weeks beginning on day 1 of cycle 1. Patients also undergo multiparametric MRI and collection of blood samples throughout the trial. Patients undergo PSMA-PET/CT scans during screening and follow up.
  Interventions: Drug: Apalutamide; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Gallium Ga 68 Gozetotide; Radiation: Guided Stereotactic Body Radiation Therapy; Procedure: Multiparametric Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PSMA-PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Other: Gallium Ga 68 Gozetotide — Undergo PSMA-PET/CT
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; AAA 517; AAA-517; AAA517; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Radiation: Guided Stereotactic Body Radiation Therapy — Undergo guided SBRT
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo multiparametric MRI
  Other Names: MP-MRI; mpMRI; Multi-parametric MRI; Multiparametric MRI
Procedure: Positron Emission Tomography — Undergo PSMA-PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial evaluates apalutamide in combination with image-guided stereotactic body radiation therapy (SBRT) for the treatment of patients with prostate cancer. Prostate cancer usually needs the hormone testosterone to grow. Apalutamide is a hormone therapy that blocks the effect of testosterone on prostate tumor cells. This may help stop the growth of tumor cells that need testosterone to grow. Image-guided SBRT is a standard treatment for some types of prostate cancer. This treatment combines imaging of cancer within the body, with the delivery of therapeutic radiation doses produced on a linear accelerator machine. SBRT uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Combining apalutamide with image-guided SBRT may increase a prostate cancer patient's chances of achieving an extremely low prostate specific antigen response, which is an early predictor of disease cure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess prostate specific antigen (PSA) complete response rates in patients with unfavorable intermediate risk prostate cancer who are receiving apalutamide monotherapy in conjunction with magnetic resonance imaging stereotactic body radiotherapy with precision dose-escalation and de-escalation to involved and uninvolved areas of the prostate, respectively.

SECONDARY OBJECTIVES:

I. Assessing time to biochemical recurrence (BCR; PSA ≥ nadir PSA + 2 ng/mL) among patients initially meeting primary endpoint.

II. Assessing patient-reported genitourinary quality of life, as assessed by the Expanded Prostate Cancer Index Composite-26 (EPIC-26) survey instrument 24 months after radiotherapy completion.

III. Assessing patient-reported bowel quality of life, as assessed by the EPIC-26 survey instrument 24 months after radiotherapy completion.

IV. Assessing radiographic persistence of disease on a prostate specific membrane antigen (PSMA) positron emission tomography/computed tomography (PET/CT) six months following hormonal therapy completion.

V. Assessing radiographic persistence of disease on a multiparametric MRI at fixed intervals (i.e., 6, 12, 18, 24, 30) months after radiotherapy completion.

VI. Assessment of longitudinal changes in patient-reported quality of life metrics on the EPIC-26 survey instrument.

VII. Physician-reported acute and late toxicities as per the Common Terminology Criteria for Adverse Events (CTCAE) scale version (v)5.0.

OUTLINE:

Patients receive apalutamide orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 or 12 months in the absence of disease progression or unacceptable toxicity. Patients undergo SBRT for 5 fractions over 1-2 weeks beginning on day 1 of cycle 1. Patients also undergo multiparametric MRI and collection of blood samples throughout the trial. Patients undergo PSMA-PET/CT scans during screening and follow up.

After completion of study treatment, patients are followed up every 3 months for up to 24 months after SBRT and then up to 60 months after SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of prostate adenocarcinoma
* Age ≥ 18
* Classified as having National Comprehensive Cancer Network unfavorable intermediate risk prostate cancer (i.e., [a] 2 of the following: PSA 10-20 ng/mL, clinical T category 2b-2c, or International Society of Urological Pathology [ISUP] grade group 2; [b] OR any 1 of [a] with ISUP grade group 3 disease; OR [c] any 1 of [a] with 50% or more cores on systematic biopsy showing prostate cancer)
* Have a Decipher genomic classifier score
* Have at least one dominant intraprostatic lesion visible on multiparametric MRI (Prostate Imaging-Reporting and Data System [PI-RADS] version 2.1 score 4 or 5)
* Have underwent a prostate specific membrane antigen (PSMA) positron emission tomography/computed tomography (PET/CT)
* Have total testosterone >= 150 ng/dL
* Adequate performance status (Eastern Cooperative Oncology Group [ECOG] 0-1)
* Hemoglobin ≥ 9.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization (at screening)
* Platelet count ≥ 100,000 x 10^9/uL independent of transfusion and/or growth factors within 3 months prior to randomization (at screening)
* Serum albumin ≥ 3.0 g/dL (at screening)
* Glomerular filtration rate (GFR) ≥ 45 mL/min (at screening)
* Serum potassium ≥ 3.5 mmol/L (at screening)
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤ 1.5 x ULN, subject may be eligible) (at screening)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 x ULN (at screening)
* Medications known to lower the seizure threshold (see list under prohibited medications) must be discontinued or substituted at least 4 weeks prior to study entry

Exclusion Criteria:

* Any evidence of spinal cord compression (radiological or clinical)
* Prior pelvic malignancy
* Prior pelvic radiation
* Concurrent malignancy other than adequately treated basal cell or squamous cell skin cancer, non-muscle invasive bladder cancer (NMIBC), or any other cancer in situ currently without evidence of recurrence or progression
* Inability to undergo radiotherapy, or hormonal therapy
* Primary small cell carcinoma of the prostate (prostate adenocarcinoma with neuroendocrine differentiation is allowed)
* Inflammatory bowel disease or active collagen vascular disease
* History of any of the following:

  * Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1 year to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign central nervous system [CNS] or meningeal disease which may require treatment with surgery or radiation therapy)
  * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization
* Current evidence of any of the following:

  * Uncontrolled hypertension
  * Gastrointestinal disorder affecting absorption
  * Known active infection (eg, human immunodeficiency virus [HIV] or viral hepatitis)
  * Any condition that in the opinion of the investigator would preclude participation in this study
  * Treatment with CYP2D6 substrates that have a narrow therapeutic index. If an alternative treatment cannot be used, a dose reduction of the CYP2D6 substrate may be considered
  * Baseline moderate and severe hepatic impairment (Child Pugh class B & C)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients achieving prostate specific antigen (PSA) of < 0.2 ng/mL | Three months after completion of apalutamide
  Will be summarized by count and percent along with the 95% confidence interval. This will then be compared to the historical control rate of 70% using a two sample z test for proportions with a one-sided p-value threshold of 0.05.

SECONDARY OUTCOMES:
Time to biochemical recurrence (BCR) | We will follow patients for five years following completion of radiotherapy. Biochemical disease status will be checked every 3 months for the first year, and every 6 months thereafter.
  Evaluated among patients initially meeting the primary endpoint. BCR is defined as PSA >= nadir PSA + 2 ng/mL. Time to BCR will be reported descriptively for each patient. Five-year biochemical recurrence free survival will be estimated by the Kaplan-Meier method as well as descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum).
Patient-reported outcomes (PROs) on the Expanded Prostate Cancer Index Composite-26 (EPIC-26) urinary domain | 24 months after completion of stereotactic body radiation therapy (SBRT)
  Changes will be analyzed with respect to whether they represent minimally important differences.
PROs on the EPIC-26 bowel domain | 24 months after completion of SBRT
  The analysis of both acute and late changes in the bowel domain of the EPIC instrument will be stratified for use of hydrogel spacers or not, as these may reduce both acute and late gastrointestinal bowel symptoms.
Radiographic persistence of disease on prostate specific membrane antigen (PSMA) positron emission tomography/computed tomography (PET/CT) | 6 months after hormonal therapy completion
  Defined by expert reader using the criterion of standardized uptake value within 20% of pre-SBRT PSMA PET/CT. Will be reported as a binary value (persistent versus not persistent).
Radiographic persistence of disease on multiparametric magnetic resonance imaging | At 6 months, 12 months, 18 months, 24 and 30 months after radiotherapy completion
  Defined by expert reader using a composite of apparent diffusion coefficient, size, and ktrans. Will be reported as a binary value (persistent vs. not persistent).
Longitudinal PROs on the EPIC-26 questionnaire in the sexual, urinary, and bowel domains | Up to 60 months
  For the EPIC-26 instrument, these will be represented by changes from baseline in the urinary incontinence, urinary obstruction, bowel, sexual function, and hormone/vitality domains. Changes will be analyzed with respect to whether they represent minimally important differences.
Physician-reported acute and late toxicities | We will follow patients for five years following completion of radiotherapy. Acute toxicity will be scored within the first 90 days after radiation. Late toxicity and patient-reported outcomes will be assessed every 3 months for the first year, and every
  Evaluated per the Common Terminology Criteria for Adverse Events scale version 5.0. Rates will be reported descriptively. The 5-year cumulative incidences of late grade ≥ 2 genitourinary and gastrointestinal toxicity will be analyzed using a cumulative incidence framework. The analysis of gastrointestinal toxicities (acute and late) will be stratified by the use of hydrogel spacers.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States